CLINICAL TRIAL: NCT01318369
Title: The Safety, Tolerability, and Analgesic Efficacy of Δ9-THC (Namisol®) in Chronic Pancreatitis Patients Suffering From Persistent Abdominal Pain
Brief Title: Efficacy Study of Δ9-THC to Treat Chronic Abdominal Pain
Acronym: Delta-pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEEL-2011-01
Record Dates: First submitted 2011-03-09; First posted 2011-03-18 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Cannabinoid; Tetrahydrocannabinol; Chronic Pancreatitis; Abdominal Pain
MeSH Terms: conditions — Pancreatitis, Chronic; Abdominal Pain | interventions — Dronabinol; Diazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Namisol (Experimental): Namisol (dronabinol) single dose 8 mg
  Interventions: Drug: Namisol
- Diazepam (Active Comparator): Diazepam single dose 5mg in subgroup non-opioid users and 10 mg in subgroup opioid users.
  Interventions: Drug: Diazepam

INTERVENTIONS:
Drug: Namisol — Single dose delta-9-tetrahydrocannabinol
  Other Names: Dronabinol; THC
  Arms: Namisol
Drug: Diazepam — Diazepam single dose 5mg in subgroup non-opioid users and 10 mg in subgroup opioid users.
  Arms: Diazepam

SUMMARY:
The main goal of this trial is to study the efficacy of Namisol® after a single dose of Δ9-THC in the treatment of pain resulting from chronic pancreatitis. Objective measures of pain processing, e.g. encephalography (EEG) and quantitative sensory testing (QST), are included to provide insight in underlying nociceptive processing.

DETAILED DESCRIPTION:
The most important symptom in chronic pancreatitis (CP) is abdominal pain. Pancreatic pain is often recurrent, intense and long-lasting, and is extremely difficult to treat. Medical analgesic therapy is considered as first choice in pain management of CP, resulting in regularly prescription of opioids. The adverse consequences of prolonged opioid use, including addiction, tolerance and opioid induced hyperalgesia, call for an alternative medical treatment. Cannabis has been used to treat pain for many centuries. Delta-9-tetrahydrocannabinol (Δ9-THC), the psychoactive substance of the cannabis plant, has been shown in previous studies to be a promising analgesic. The development of Namisol®, a tablet containing purified Δ9-THC showing an improved and reliable pharmacokinetic profile, provides the opportunity to test the analgesic potential of Δ9-THC in favourable conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patient has chronic pancreatitis, diagnosed using the Marseille and Cambridge Classification System (addendum II).37
* Patient suffers from chronic abdominal pain typical for pancreatitis, meet the criteria for chronic pain according ISAP (intermittent or persistent pain on a daily basis in at least 3 months)38, and consider their pain must as severe enough for medical treatment (average NRS ≥ 3).
* Patient in the opioid group takes stable doses of opioids, e.g. morphine or tramadol, for the past 2 months on the day of screening. Stable dose intake is defined as a daily equivalent sum of opioid intake according medical prescription within a small deviation range as judged by the (principal) investigator.
* Patient in the non-opioid group does not take any opioids for the past 2 months on the day of screening.

Exclusion Criteria:

* Patient used any cannabinoid (by smoking cannabis or oral intake) for at least one year on the day of screening.
* Patient does not feel a pinprick test in the lower extremities, due to affected sensory input (e.g. neuropathy as a result of diabetes mellitus).
* Patient has a body mass index (BMI) below 18 or above 31.2 kg/m2.
* Patient suffers from serious painful conditions other than chronic pancreatitis or had any major pre-existing chronic pain syndrome.
* Patient has a (history of) a significant medical disorder that, in the opinion of the investigator, may interfere with the study or may pose a risk for the patient.
* Patient uses any kind of concomitant medication that, in the opinion of the investigator, may interfere with the study or may pose a risk for the patient (e.g. HIV antivirals).
* Patient takes amitriptyline on a daily basis.
* Patient takes more than 20 mg benzodiazepines 6 hours prior or following intake of study medication (11 hour am) according prescription.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Pain intensity (VAS pain) | Repeatedly; baseline until 6 hours after administration
  Pain intensity (VAS pain at rest and on movement)

SECONDARY OUTCOMES:
EEG | Repeatedly; baseline until 6 hours after administration
  Spontaneous EEG and evoked potentials to noxious electrical stimuli
QST | Repeatedly; baseline until 6 hours after administration
  Quantitative Sensory Testing, using pressure pain tolerance and electrical thresholds
Body sway | Repeatedly; baseline until 6 hours after administration
  Static body sway

CONTACTS AND LOCATIONS:
Overall Officials: Harry van Goor, MD PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands